CLINICAL TRIAL: NCT06093997
Title: Study on the Treatment of Cervical Spondylosis of Qi Stagnation and Blood-stasis Type by Moving Cupping Combined with Bloodletting
Brief Title: Study on the Treatment of C/S of Qi Stagnation and Blood-stasis Type by Moving Cupping with Bloodletting
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Gao Mingli, Attending Doctor, Shanghai University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: I111
Record Dates: First submitted 2023-09-20; First posted 2023-10-23 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Cervical Spondylosis
Keywords: Cervical Spondylosis of Qi Stagnation and Blood-stasis Type
MeSH Terms: conditions — Spondylosis | interventions — Cupping Therapy; Bloodletting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Cupping and bloodletting therapy
  Interventions: Other: Cupping; Other: Bloodletting
- Control Group (Experimental): Massage treatment
  Interventions: Other: Massage treatment

INTERVENTIONS:
Other: Massage treatment — The patient sits upright and the neck naturally relaxes. The doctor uses techniques such as pressing and kneading to relax the soft tissues of the neck, and massages points such as FengMen, FengChi, JingJiaji, JianJing,Tianzong and so on. The focus is on using muscle relaxation techniques around the soft tissues of spasms and pain areas to relax the patient's neck and shoulders. All procedures were performed from mild to severe, once a week for 15 minutes each time, for a total of 4 weeks of treatment.
  Arms: Control Group
Other: Cupping — Use a 4-5cm diameter suction cupping for cupping. The treatment area is coated with glycerol, and the cupping is aspirated and adsorbed on the skin. The cupping is slowly pushed along the patient's neck, along the urinary bladder channel of Foot-Taiyang and governor's meridians from top to bottom, repeating back and forth 9 times. Once a week, for a total of 4 weeks of treatment.
  Arms: Experimental Group
Other: Bloodletting — the doctor takes JianZhongShu, one on the left and one on the right, with a total of 2 acupoints. After disinfecting with 75% alcohol cotton balls, the patient is quickly pricked 5 times with a blood collection needle, and cupping is performed at the needle hole. After 5 minutes, remove the jar, wipe the blood clean, and disinfect the needle hole. Once a week, for a total of 4 weeks of treatment.
  Arms: Experimental Group

SUMMARY:
The goal of this Clinical randomized controlled trial is to evaluate the therapeutic effect of cupping combined with bloodletting in the treatment of cervical spondylosis of qi stagnation and blood stasis type. The main question it aims to answer is: How to remove stasis and prolong the time of promoting blood circulation. Participants will adopt the combination of cupping and bloodletting therapy.Researchers will compare massage treatment to see if the combination of cupping and bloodletting puncture is more effective in treating cervical spondylosis of qi stagnation and blood stasis type

DETAILED DESCRIPTION:
In recent years, the incidence rate of cervical spondylosis has continued to rise. Among them, cervical spondylosis of qi stagnation and blood stasis type, mainly characterized by neck and shoulder pain, is mainly treated by activating blood to remove blood stasis, regulating qi and unblocking collaterals due to blood stasis and qi stagnation and blocked muscles and collaterals. Massage therapy is the most commonly used in clinical practice, but its maintenance time is short and clinical symptoms recur. How to remove stasis and prolong the time of blood circulation is the key to treatment.

Walking cupping has the function of unblocking meridians and regulating qi and blood. Compared to massage, kneading, and pressing to stimulate acupoints, walking cupping also increases the scope of stimulation. If it is not clear, it will cause pain, while if it is clear, it will not cause pain. By pricking the meridians and releasing blood, it can activate the meridians, dispel blood stasis, and relieve pain. After cupping, pricking and bleeding can increase the amount of bleeding. The combination of the two can further alleviate symptoms such as neck and shoulder pain and stiffness in patients, and improve the therapeutic effect.

Based on this, this project randomly divided 62 patients with cervical spondylosis of qi stagnation and blood stasis type into a control group and an experimental group. The control group received massage treatment, while the experimental group received cupping combined with bloodletting therapy. Using the Northwick Park Neck Pain Scale score as the primary outcome measure; Cervical mobility measurement, traditional Chinese medicine syndrome score, and adverse reactions are secondary outcome indicators. Objectively evaluate the efficacy of cupping combined with bloodletting puncture in the treatment of cervical spondylosis patients with qi stagnation and blood stasis, promote suitable techniques with traditional Chinese medicine characteristics for treating cervical spondylosis, and help cervical spondylosis patients recover their daily life and work abilities as soon as possible.

ELIGIBILITY:
Inclusion criteria

* Patients who meet the diagnostic criteria (Traditional Chinese medicine diagnosis conforms to the diagnostic criteria for cervical spondylosis of qi and blood stasis type in the "Guiding Principles for Clinical Research of Traditional Chinese Medicine New Drugs". Western medicine diagnosis adopts the diagnostic criteria for cervical spondylosis developed at the "Third National Symposium on Cervical Spondylosis" held in April 2008 at Dongfang Hospital Affiliated to Tongji University.);

  * The course of the disease is more than 3 months;

    * Gender unlimited ④ Age 18-80 years old; ⑤ No history of neck and shoulder surgery; ⑥ Those who have not received relevant treatment in the past month; ⑦ Those who voluntarily participate in this study and sign an informed consent form.

Exclusion criteria

* Head and neck injuries;

  * Patients with a tendency to bleed;

    * Pregnant and lactating women;

      * Concomitant with serious primary diseases such as heart, cerebrovascular disease, liver, kidney, etc;

        * Individuals with severe mental illness or cognitive impairment;

          * Individuals with acute infection or local skin damage due to local trauma; ⑦ Patients with infectious diseases transmitted through blood; ⑧ Those who cannot persist in receiving treatment according to the prescribed time.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The Northwick Park Neck Pain Questionnaire | Before treatment, 1 week after treatment, 4 weeks after treatment, and 1 month after the end of treatment
  Including clinical symptoms (degree and duration of neck pain, etc.) and quality of life (sleep time, impact on reading and watching TV, impact on social activities, etc.), a total of 9 items, with a total score of 32-36 points. The final score is converted into a percentage system, and the higher the score, the worse the cervical condition.

SECONDARY OUTCOMES:
Measurement of cervical spine mobility | Before treatment, 1 week after treatment, 4 weeks after treatment, and 1 month after the end of treatment
  Measure the angles of cervical spine flexion, extension, left flexion, right flexion, left rotation, and right rotation using a cervical spine mobility measuring instrument.
Scoring of Traditional Chinese Medicine Syndrome | Before treatment, 1 week after treatment, 4 weeks after treatment, and 1 month after the end of treatment
  Referring to the Guiding Principles for Clinical Research of New Chinese Medicine (Trial), the symptom grading of cervical spondylosis includes strong neck pain, limb numbness, dizziness, headache, limb paralysis, palpitations, insomnia, tinnitus, and chills; Score 0, 2, 4, and 6 points based on none, light, medium, and heavy, respectively. The total score is 0-54 points, and the lower the total score, the lighter the clinical symptoms.
Adverse reactions | Before treatment, 1 week after treatment, 4 weeks after treatment, and 1 month after the end of treatment
  Record the occurrence of adverse events during the patient's treatment, including the type and number of adverse reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Xu, chief, Study Director — Shanghai Qigong Institute
Locations (1):
- Medical Outpatient Department of Shanghai Qigong Research Institute, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
This plan has not been approved by the Clinical Ethics Committee.

REFERENCES:
- [Background] Cervical Spondylosis Professional Committee of the Chinese Rehabilitation. Medical Association Guidelines for Diagnosis, Treatment and Rehabilitation of Cervical Spondylosis [S]: Beijing: Cervical Spondylosis Professional Committee of the Chinese Rehabilitation Medical Association, 2010.
- [Background] Jin Y. The clinical research progress of traditional Chinese medicine characteristic therapy in the treatment of cervical spondylosis. Chinese folk therapy. 2017. 25 (09): 103-104.
- [Background] Lian L, Zhang S. Clinical observation on the treatment of vertebral artery type cervical spondylosis with heat sensitive moxibustion combined with bloodletting. Journal of Modern Integrated Traditional Chinese and Western Medicine. 2018. 27 (31): 3468-3470.
- [Background] Chen L, Li M, Fan L, Zhu X, Liu J, Li H, Xu Z, Chen J, Liang Z, Liu Z, Feng L, Chen X, He Q, Chen X, Ou A, He J, Ma R, Ning B, Jiang L, Li S, Fu W. Optimized acupuncture treatment (acupuncture and intradermal needling) for cervical spondylosis-related neck pain: a multicenter randomized controlled trial. Pain. 2021 Mar 1;162(3):728-739. doi: 10.1097/j.pain.0000000000002071. PMID 32947547
- [Background] Wu P, Wang J, Wang W, Gu J, Wu Z. Study on the Optimization of Acupuncture and Bleeding Analgesia Schemes for Cervical Spondylosis of Qi Stagnation and Blood Stasis Type. Chinese Journal of Basic Traditional Chinese Medicine. 2018. 24 (11): 1582-1585.
- [Background] Hai Q, Zhao L. Clinical observation on the treatment of cervical spondylosis of vertebral artery type with cupping and bloodletting therapy of Mongolian medicine combined with acupuncture and moxibustion. Chinese Journal of Ethnic Medicine. 2020.26 (08): 28-29.
- [Background] Yang X. Observation on therapeutic effect of Chinese massage combined with acupuncture and moxibustion on cervical spondylotic radiculopathy. Chinese folk therapy. 2014. 22 (07): 26.
- [Background] Luo G, Tang Z. Observation on the therapeutic effect of moving cupping combined with stasis needle technique on lumbar fasciitis. Journal of Practical Traditional Chinese Medicine. 2015. 31 (11): 1044.
- [Background] Jiang Q. The combination of cupping and scraping for the treatment of back myofasciitis. Massage and Rehabilitation Medicine June. 2015 (21): 18-19.
- [Background] Peng T, Gong H, Hu S, Zhou C, Xie G, Xiong J. Clinical observation on the treatment of neck shoulder syndrome with scraping combined with cupping therapy. Shanghai acupuncture and moxibustion Journal. 2016. 35 (06): 713-715.
- [Background] Jiang M, Peng T. The combination of meridian scraping and cupping therapy for the treatment of neck dorsalis myofascitis. Journal of Traditional Chinese Medicine. 2022. 37 (01): 197-200.
- [Background] Li H, Ma F, Zhang W, Zhao N, Hai X, Wang J. Clinical study on the treatment of nerve root cervical spondylosis of qi stagnation and blood stasis type with phased differentiation and massage therapy. Chinese Journal of Traditional Chinese Medicine. 2017. 35 (04): 939-942.
- [Background] Hu Y, Yang J, Li L. Progress in the treatment of vertebral artery type cervical spondylosis with acupuncture, moxibustion and massage. Hebei Medicine. 2015. 21 (08): 1532-1534.
- [Background] Ma Z, Fu A, Wang Y, Chen Z. The therapeutic effect of acupuncture combined with bloodletting therapy on cervical spondylotic radiculopathy and its impact on pain and blood viscosity. National Medical Forum. 2019. 34 (01): 23-24.
- [Background] Huang F, Wang H, Sun C, Wang L, Yin J, Zhang Q. Acupuncture and push combined with bloodletting therapy for treating 35 cases of cervical spondylosis with qi stagnation and blood stasis. Liaoning Journal of Traditional Chinese Medicine. 2019. 46 (01): 144-147.
- [Background] Peng T, Wan G, Shan R. Scraping combined with cupping for the treatment of 180 cases of neck shoulder syndrome. Modern Distance Education of Traditional Chinese Medicine in China. 2014. 12(07): 68-69.
- [Background] Leak AM, Cooper J, Dyer S, Williams KA, Turner-Stokes L, Frank AO. The Northwick Park Neck Pain Questionnaire, devised to measure neck pain and disability. Br J Rheumatol. 1994 May;33(5):469-74. doi: 10.1093/rheumatology/33.5.469. PMID 8173853